CLINICAL TRIAL: NCT03743116
Title: Incidence of Postoperative Orthostatic Intolerance and Postoperative Orthostatic Hypotension in Patients Undergoing Unilateral Total Knee Arthroplasty
Brief Title: Postoperative Orthostatic Intolerance and Hypotension in Unilateral TKA
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Kehlet, Henrik, M.D., Ph.D. (Individual)
Responsible Party: Principal Investigator, Ana-Marija Hristovska, Principal Investigator, Medical Doctor, Hvidovre University Hospital
Other Study IDs: H-18049929
Record Dates: First submitted 2018-11-08; First posted 2018-11-15 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Orthostatic Intolerance; Orthostatic Hypotension; Postoperative Complications
Keywords: Orthostatic Intolerance; Orthostatic Hypotension; Knee arthroplasty
MeSH Terms: conditions — Orthostatic Intolerance; Hypotension, Orthostatic; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Orthostatic intolerant (OI): Patients that experience symptoms of orthostatic intolerance (dizziness, nausea, vomiting, blurry vision or syncope) or orthostatic hypotension (fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg) during mobilisation
- Orthostatic tolerant (OT): Patients that do not experience symptoms of orthostatic intolerance (dizziness, nausea, vomiting, blurry vision or syncope) or orthostatic hypotension (fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg) during mobilisation

SUMMARY:
Incidence of Postoperative Orthostatic Intolerance and Postoperative Orthostatic Hypotension in Patients Undergoing Unilateral Total Knee Arthroplasty

DETAILED DESCRIPTION:
Early postoperative mobilization is a cornerstone in the so-called fast track multimodal perioperative approach and is essential in preventing postoperative morbidity and reducing hospital length-of-stay. Intact orthostatic blood pressure regulation is essential for early postoperative mobilization. However, early postoperative mobilization can be delayed due to postoperative orthostatic hypotension (POH) defined as a fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg or due to postoperative orthostatic intolerance (POI), characterized by dizziness, nausea, vomiting, blurred vision or syncope during mobilization.

Previous prospective studies of major surgery have reported that OI and OH are common problem during early postoperative mobilization, with a prevalence of 42-50%. Retrospective studies with a less-defined mobilization protocols have reported am OI prevalence in the range of 12-60 % across surgical procedures.

The aim of our study is to determine the incidence of OI during early postoperative mobilization in fast track unilateral total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Written informed consent
* Patients that speak and understand Danish
* Patients undergoing primary unilateral total knee arthroplasty in spinal anesthesia and standardized fast-track setting

Exclusion Criteria:

* Alcohol or drug abuse
* Cognitive dysfunction
* Known orthostatic hypotension
* Use of anxiolytic drugs

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary unilateral total knee arthroplasty in spinal anesthesia and standardized fast-track setting
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of orthostatic intolerance | 6 hours postoperatively
  Symptoms of orthostatic intolerance: dizziness, nausea, vomiting, blurry vision or syncope during mobilization
Incidence of orthostatic hypotension | 6 hours postoperatively
  Orthostatic hypotension is defined as a fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg during mobilization

SECONDARY OUTCOMES:
Changes in systolic arterial pressure (SAP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg
Changes in diastolic arterial pressure (DAP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg
Changes in mean arterial pressure (MAP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg
Changes in systemic vascular resistance (SVR) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg⋅min⋅mL-1
Changes in cardiac output (CO) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL/min
Changes in stroke volume (SV) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Marija Hristovska, MD, Principal Investigator — Department of Anesthesiology, Hvidovre Hospital, Copenhagen
Locations (1):
- Hvidovre University Hosptial, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No